CLINICAL TRIAL: NCT03234985
Title: Study of Intracellular Nucleotide Pools Determination as Biomarker of the Efficacy of the Induction Treatment in Acute Myeloid Leukemia
Acronym: NUCLARA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0351
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute myeloid leukemia patients: Patients over 18 years with acute myeloid leukemia
  Interventions: Biological: Biological analyses

INTERVENTIONS:
Biological: Biological analyses — Biological analyses will be realized on samples collected before induction treatment and at the end of bone marrow aplasia i.e. about day 30 to determine the nucleotide pools in peripheral blood mononuclear cells.

SUMMARY:
Treatment of acute myeloid leukemia (AML) consists in two main phases: induction and consolidation. Standard chemotherapy combination for induction treatment associates cytarabine (AraC), a nucleoside analog, and an anthracycline (most often daunorubucin). About 60-70% of patients achieved complete remission after this standard chemotherapy. As cytarabine competes with endogenous nucleotides to exert its activity, the aim of this protocol is to study in vivo the effect of intracellular nucleotide pools on the efficacy of the induction treatment. Thus, intracellular nucleotides levels will be determined in peripheral blood mononuclear cells of patients with acute myeloid leukemia before treatment, and results will be compared with the efficacy of the treatment. This parameter will be assessed by the achievement of complete remission.

ELIGIBILITY:
Patients Inclusion Criteria:

* age over 18 years
* acute myeloid leukemia
* standard induction chemotherapy with cytarabine and daunorubicin
* patients who received the information and did not object to participate to the study

Patients Exclusion Criteria:

- patients with acute myeloid leukemia 3

healthy volunteers Inclusion Criteria :

* adults without known hematological disease,
* adults who received the information and did not object to participate in the study

healthy volunteers Exclusion Criteria :

- Volunteers with known hematological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients or healthy volunteers over 18 years with acute myeloid leukemia (except acute myeloid leukemia3)
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Complete remission | 30 days
  Primary endpoint will be the achievement of complete remission after induction treatment and bone marrow aplasia.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hématologie - Centre Hospitalier Lyon Sud - Hospices Civils de LYON, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No